CLINICAL TRIAL: NCT03958383
Title: Phase I/II Intratumoral Administration of Hu14.18-IL2, With Local Radiation, Nivolumab and Ipilimumab in Subjects With Advanced Melanoma
Brief Title: IT-hu14.18-IL2 With Radiation, Nivolumab and Ipilimumab for Melanoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry); AnYxis Immuno-Oncology GmbH (Unknown); Provenance Biopharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW16134; 2017-1464 (Other: Institutional Review Board); R35CA197078 (NIH); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 7/30/2020 (Other: UW Madison)
Record Dates: First submitted 2019-05-07; First posted 2019-05-22 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — lorukafusp alfa; Radiotherapy; Nivolumab; spartalizumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation design to determine maximum tolerated dose / maximum administered dose for each of 4 cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Groups (Experimental): PHASE IA: As described above. Participants receive hu14.18-IL2 fusion protein intratumorally (IT).
  PHASE IB: As described above. Participants undergo palliative RT and hu14.18-IL2 fusion protein IT as in phase IA.
  PHASE IC: As described above. Participants undergo palliative RT, receive nivolumab, and hu14.18-IL2 fusion protein IT as in phase IA.
  PHASE ID: As described above. Participants undergo palliative RT, receive nivolumab in combination with ipilimumab, and hu14.18-IL2 fusion protein IT as in phase IA.
  Interventions: Biological: hu14.18-IL2; Radiation: Radiation Therapy; Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: hu14.18-IL2 — A recombinant fusion protein linking the monoclonal antibody (mAb) hu14.18 with interleukin-2 (IL2), administered IT
  Other Names: immunocytokine
Radiation: Radiation Therapy — Palliative radiation therapy
  Other Names: Radiotherapy
Biological: Nivolumab — Human programmed death receptor (PD-1) blocking antibody, given IV
  Other Names: anti-PD-1
Biological: Ipilimumab — Monoclinal antibody that targets cytoxic T-lymphocyte-associated protein 4 (CTLA-4), given IV
  Other Names: anti-CTLA-4

SUMMARY:
This phase I/II trial is designed to determine the maximum tolerated dose or the maximum administered dose of intratumoral administration of hu14.18-IL2 and to evaluate side effects of intratumoral hu14.18-IL2 when given alone, after radiation therapy, after radiation therapy and in combination with nivolumab, and after radiation therapy and in combination with nivolumab and ipilimumab in patients with melanoma that is advanced (stage IV) or with melanoma that cannot be removed by surgery and is considered surgically incurable. Hu14.18-IL2 is a molecule called a fusion protein that can bind to some tumor cells and cause immune cells to become activated to kill tumor cells. Radiation therapy is a type of cancer treatment that uses beams of high energy x-rays to kill tumor cells and shrink tumors. Immunotherapy with immune checkpoint inhibitors, such as nivolumab and ipilimumab, can help the body's immune system attack cancer by releasing the "brakes" on the immune system to allow cancer fighting immune cells to remain activated. This study will evaluate whether giving intratumoral hu14.18-IL2 with radiation therapy, nivolumab and ipilimumab has antitumor activity for participants with advanced melanoma.

After completion of study treatment, participants are followed up at 30 days, every 12 weeks for up to 2 years, and then every 6 months thereafter.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) of intratumoral (IT)-Hu14.18-IL2 fusion protein (hu14.18-IL2) in subjects with advanced melanoma (Phase IA)

II. Evaluate the safety and tolerability of IT-hu14.18-IL2 when given alone (Phase IA)

III. Determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) of IT-hu14.18-IL2 after receiving palliative radiation therapy (RT) in subjects with advanced melanoma (Phase IB)

IV. Evaluate the safety and tolerability of the combination of palliative RT with IT-hu14.18-IL2 (Phase IB)

V. Determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) of IT-hu14.18-IL2 after receiving palliative RT and in combination with nivolumab in subjects with advanced melanoma (Phase IC)

VI. Evaluate the safety and tolerability of the combination of palliative RT, nivolumab and IT-hu14.18-IL2 (Phase IC)

VII. Determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) of IT-hu14.18-IL2 after receiving palliative RT and in combination with nivolumab and ipilimumab in subjects with advanced melanoma (Phase ID)

VIII. Evaluate the safety and tolerability of the combination of palliative RT, nivolumab, ipilimumab and IT-hu14.18-IL2 (Phase ID)

IX. Evaluate local and systemic objective tumor responses to treatment with IT-hu14.18-IL2 in combination with palliative RT, nivolumab, and ipilimumab (Phase ID)

SECONDARY OBJECTIVES:

I. Evaluate progression-free survival (PFS), overall survival (OS), clinical benefit (CB, defined as complete response (CR) + partial response (PR) + stable disease (SD)) and duration of response to hu14.18-IL2 in combination with RT, nivolumab and ipilimumab.

II. Evaluate pathologic (tissue) evidence of immune response at the injection site and untreated sites.

III. Evaluate PFS, CB and duration of response to hu14.18-IL2 in combination with palliative RT, nivolumab and ipilimumab based on resistance to prior treatment with anti-CTLA-4 and/or anti PD1/PD-L1 antibody.

IV. Evaluate serial serum samples to determine the pharmacokinetics of hu14.18-IL2 administered intratumorally.

V. Evaluate each subject's tumor cells for expression of GD2 and PD-L1, and determine if either antitumor activity or selected treatment-associated biologic effects are more likely for tumors that are GD2+ then GD2- and PD-L1+ than PD-L1-.

VI. Evaluate whether PD-L1 expression is induced or augmented from baseline following initiation of treatment (by comparing serial biopsies).

VII. Evaluate the immunologic activation induced in vivo by IT-hu14.18-IL2, addressed by in vitro cellular, serologic and flow cytometry immune assays.

VIII. Evaluate for histological evidence of antitumor activity based on the presence of necrotic tumor cells, inflammatory infiltrate, cellular phenotype of infiltrate, and presence of hu14.18-IL2 within the tumor at selected post-treatment timepoints.

IX. Evaluate circulating tumor cells, exosomes, endogenous antibodies, and/or deoxyribonucleic acid (DNA) as exploratory biomarkers associated with clinical response to IT-hu14.18-IL2 in combination with RT, nivolumab and ipilimumab.

X. Evaluate serial peripheral blood mononuclear cell (PBMC) samples to monitor the induction of T cell responses to melanoma-associated antigens.

XI. Evaluate objective tumor responses, both locally and systemically (by immune-related response criteria), in Phases IA, IB and IC of this trial (involving IT-hu14.18-IL2 alone and in combinations with palliative RT, and with palliative RT and nivolumab, respectively).

OUTLINE: This is a dose escalation study of hu14.18-IL2 fusion protein.

PHASE IA: Participants receive hu14.18-IL2 fusion protein intratumorally (IT) once daily (QD) on days 1-3. Treatment repeats every 21 days for cycles 1-4. Participants who are eligible may continue to receive hu14.18-IL2 fusion protein maintenance therapy QD on days 1-3 beginning with cycle 5. Maintenance cycles repeat every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. A total of 9-18 participants will be enrolled in 3 escalating dose levels to determine the Maximum Tolerated Dose (MTD)/Maximum Administered Dose (MAD) of hu14.18-IL2 in Phase IA.

PHASE IB: Participants undergo palliative RT on days -8 to -4 of cycle 1 only. Participants also receive hu14.18-IL2 fusion protein IT as in phase IA. Treatment with hu14.18-IL2 repeats every 21 days for cycles 1-4. Participants who are eligible may continue to receive hu14.18-IL2 fusion protein maintenance therapy QD on days 1-3 beginning with cycle 5. Maintenance cycles repeat every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. The MTD/MAD of IT-hu14.18-IL2 following palliative RT will be determined starting 1 dose level below the Phase IA determined MTD/MAD of IT-hu14.18-IL2 up to the Phase IA determined MTD/MAD.

PHASE IC: Participants undergo palliative RT on days -8 to -4 of cycle 1 only. Nivolumab (3 mg/kg) is given every 2 weeks for up to 1 year with the initial dose given between day -7 and day -1 of cycle 1. Participants also receive hu14.18-IL2 fusion protein IT as in phase IA. Treatment with hu14.18-IL2 repeats every 21 days for cycles 1-4. Participants who are eligible may continue to receive hu14.18-IL2 fusion protein maintenance therapy QD on days 1-3 beginning with cycle 5. Maintenance cycles repeat every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. The MTD/MAD of IT-hu14.18-IL2 following palliative RT in combination with nivolumab will be determined starting 1 dose level below the Phase IB determined MTD/MAD of IT-hu14.18-IL2 up to the Phase IB determined MTD/MAD.

PHASE ID: Participants undergo palliative RT on days -8 to -4 of cycle 1 only. Nivolumab (1 mg/kg) in combination with ipilimumab (3 mg/kg) is given every 3 weeks for 4 cycles with the initial dose given between day -7 and day -1 of cycle 1. Following 4 cycles, no additional ipilimumab will be administered. Following cycle 4, maintenance nivolumab (3 mg/kg) can be given for up to one year. Participants also receive hu14.18-IL2 fusion protein IT as in phase IA. Treatment with hu14.18-IL2 repeats every 21 days for cycles 1-4. Participants who are eligible may continue to receive hu14.18-IL2 fusion protein maintenance therapy QD on days 1-3 beginning with cycle 5. Maintenance cycles repeat every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. The MTD/MAD of IT-hu14.18-IL2 following palliative RT in combination with nivolumab and ipilimumab will be determined starting 1 dose level below the Phase IC determined MTD/MAD of IT-hu14.18-IL2 up to the Phase IC determined MTD/MAD. A total of 28 participants will be enrolled at the Phase ID MTD/MAD of IT-hu14.18-IL2.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically proven, malignant melanoma, that is advanced (stage IV) or is unresectable and therefore considered surgically incurable
* Subject's disease must be measurable by immune-related RECIST criteria using clinical assessments or imaging
* Subjects must have at least one (1), but preferably two (2), sites of readily accessible, superficial disease (i.e., cutaneous, subcutaneous, and/or readily-palpable lymphadenopathy) that are amenable to repeated hu14.18-IL2 injections and two (2) to four (4) biopsies (designated Lesions A (index lesion) and B). These lesions must be at least 1 cm, but no greater than 5 cm, in longest diameter.

  * If there are two lesions, one will be injected with hu14.18-IL2 and undergo biopsies. The second will not undergo injections with hu14.18-IL2, but will undergo two biopsies and be observed clinically. It is preferable, but not required, that these lesions have not received prior RT.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Subjects must have received or declined at least one FDA approved immunotherapy treatment demonstrating an impact on survival (i.e: anti-CTLA-4 antibody, anti-PD-1 antibody, IL2, etc).
* Subjects with Central Nervous System (CNS) metastases are eligible if the CNS lesions are stable for at least 2 months and if tapered off treatment doses of systemic corticosteroids for at least 2 weeks prior to enrollment on the trial. Management with maintenance physiologic doses of corticosteroids is acceptable.
* Subjects to be entered into Phase IB, IC and ID must be evaluated by a radiation oncologist and determined to have a need for palliative RT based on current or imminent symptoms at a tumor site that is also injectable. If palliative RT is needed to one or more disease sites, a separate site of disease that does not require RT must remain to enable assessment of systemic disease response.
* Subjects must have adequate bone marrow, liver, and renal function as defined by:

  * Total White Blood Cell (WBC) > 3,000/mm3 (or total neutrophil count > 1,500/mm3), platelets >100,000/mm3, and hemoglobin > 10 g/dL.
  * AST/ALT ≤ 3 x the upper limit of normal. Total bilirubin ≤ 1.5 x the upper limit of normal (< 3.0 mg/dL for subjects with Gilbert's Syndrome).
  * Serum creatinine ≤ 1.5 x the upper limit of normal
* Subjects with a history of ischemic cardiac disease must complete a stress radionuclide scan with results that show no evidence of myocardial ischemia or heart failure, as well as normal pulmonary function
* Subjects must be willing and able to provide informed written consent for the study.
* Subjects must have no immediate requirements for palliative chemotherapy, or surgery. Subjects in Arm 1A must have no immediate requirement for palliative RT.
* Subjects must be willing and able to discontinue antihypertensive medications if advised to do so for the days of hu14.18-IL2 administration.
* Subjects must have a washout period of at least 28 days between any prior systemic anti-cancer therapy (including immunotherapies) and the first dose of study drug(s).

Exclusion Criteria:

* Subjects with a diagnosed auto-immune disease (exceptions: subjects with controlled diabetes mellitus type I, thyroid disease, vitiligo and alopecia areata not requiring treatment with immunosuppressants are eligible)

  * Subjects with a history of diabetes mellitus requiring systemic therapy within the past 3 months (i.e. either oral hypoglycemic agents or insulin) must have a documented Hemoglobin A1c <8.0% at the time of enrollment.
* Subjects with known genetic conditions causing pre-disposition to RT toxicity (i.e: Li-Fraumeni, ATM deficiency, active scleroderma, etc).
* Subjects who cannot provide independent, legal, informed consent.
* Women of childbearing potential will be excluded if they are pregnant, nursing, or not willing to use effective contraception, as discussed with the treating physician, during the treatment period. A negative pregnancy test (serum or urine) is required for women of child bearing potential within 14 days before study registration.

  * A person of childbearing potential is anyone (regardless of sexual orientation, gender identity, having undergone tubal ligation, or remaining celibate by choice) who was born with a uterus and at least one ovary and meets the following criteria

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had a menses at any time in the preceding 12 consecutive months).
* Subjects with symptoms of ischemic cardiac disease, congestive heart failure, or myocardial infarction within the immediate preceding 6 months and/or uncontrolled cardiac rhythm disturbance
* Subjects with significant psychiatric disabilities or seizure disorders
* Subjects with symptomatic pleural effusions or ascites.
* Subjects with organ allografts
* Subjects who require, or are likely to require, systemic treatment doses of corticosteroids, or other immunosuppressive drugs, or have used them within 2 weeks of registration (clarification: subjects receiving physiologic maintenance or replacement doses of systemic steroids are eligible).
* Subjects with significant intercurrent illnesses per physician discretion.
* Subjects with active or acute infections or active peptic ulcers, unless these conditions are adequately corrected or controlled, in the opinion of the treating physician.
* Subjects with a second malignancy other than adequately treated non-melanoma skin cancer. Subjects will be considered eligible if they have been continuously disease free for > 5 years from a second malignancy prior to the time of enrollment.
* Subjects with known human immunodeficiency virus (HIV) infection, active or chronic hepatitis B or hepatitis C infection, or with clinical evidence of hepatitis.
* Subjects with a clinically significant neurologic deficit or objective peripheral neuropathy (Grade ≥2).
* Subjects with known hypersensitivity to hu14.18-IL2 or human immunoglobulin, or those who experienced significant immune-related adverse events requiring treatment with steroids or other immunosuppressant therapy during prior treatment with ipilimumab, or anti-PD1/PD-L1 checkpoint blockade therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | up to 2 years
  The number and severity of toxicity incidents per (Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 will be summarized with frequency and proportion. The 95% confidence interval for the proportion of subjects with severe complications (grade 3 or higher toxicities) will be constructed.
Maximum Tolerated Dose (MTD) | up to 21 days
  The MTD is defined as the highest dose level at which less than 33% of the subjects experience a Dose Limiting Toxicity (DLT). DLT will be defined as grade 3 or 4 toxicity that is possibly, probably or definitely related to IT-hu14.18-IL2 graded according to CTCAE v. 5.0. A standard 3+3 design and descriptive statistics will primarily be generated to summarize the data.
Maximum Administered Dose (MAD) | up to 21 days
  The MAD is defined as the highest safely tolerated dose where less than 33% subjects experience a DLT but no higher dose level has been assessed. Descriptive statistics will primarily be generated to summarize the data.

SECONDARY OUTCOMES:
Objective Tumor Response (OR) | Up to 5 years
  OR will be summarized using descriptive statistics. Furthermore, a point estimate along with the 95% confidence interval for the proportion of subjects with OR will be provided. Clinical outcome of OR will be summarized by dose level for Phase IC.
Progression Free Survival (PFS) | Up to 5 years
  The length of time from the start of treatment until disease progression or death. Kaplan-Meier method will be used to estimate the survival distribution of progression-free survival for the Phase ID expansion cohort.
Overall Survival (OS) | Up to 5 years
  The length of time from the start of treatment until death from any cause. Kaplan-Meier method will be used to estimate the survival distribution of overall survival for the Phase ID expansion cohort.
Clinical Benefit (CB) | Up to 5 years
  The status of achieving complete response, partial response or stable disease in response to treatment. Clinical Benefit will be summarized using descriptive statistics. Furthermore, a point estimate along with the 95% confidence interval for the proportion of subjects with clinical benefit will be provided.
Duration of Response | Up to 5 years
  The length of time from documentation of tumor response until disease progression. Kaplan-Meier method will be used to estimate the survival distribution for the Phase ID expansion cohort.
Immunologic Parameters: Change in Antibody Dependent Cell-Mediated Toxicity (ADCC) Function | Baseline, Cycle 3 day 1, Cycle 5 day 1, End of Treatment (up to 13 cycles) (cycles 1-4 are 21 days, 5+ are 28 days)
  Immunologic activation induced in vivo by intratumoral (IT)-hu14.18-IL2 fusion protein will be evaluated using both in vivo and in vitro analyses. Changes between assessment time points will be evaluated using a paired t-test or non-parametric Wilcoxon signed rank test, depending on the scale and distribution of the endpoint.
Immunologic Parameters: Change in Natural Killer (NK) Cell Function | Baseline, Cycle 3 day 1, Cycle 5 day 1, End of Treatment (up to 13 cycles) (cycles 1-4 are 21 days, 5+ are 28 days)
  Immunologic activation induced in vivo by intratumoral (IT)-hu14.18-IL2 fusion protein will be evaluated using both in vivo and in vitro analyses. Changes between assessment time points will be evaluated using a paired t-test or non-parametric Wilcoxon signed rank test, depending on the scale and distribution of the endpoint.
Immunologic Parameters: Change in Soluble Interleukin-2 Receptor alpha (IL-2 alpha) Levels | Baseline; Cycle 1 days 1,4,8; Cycle 4 days 1,4,8; Cycle 7 days 1,4,8; Cycle 10 day 1,4,8 (cycles 1-4 are 21 days, 5+ are 28 days)
  Immunologic activation induced in vivo by intratumoral (IT)-hu14.18-IL2 fusion protein will be evaluated using both in vivo and in vitro analyses. Changes between assessment time points will be evaluated using a paired t-test or non-parametric Wilcoxon signed rank test, depending on the scale and distribution of the endpoint.
Histological Parameters: Change in Necrotic Tumor Cells from Baseline | Baseline, Cycle 1, Cycle 2, Cycle 4 (cycles 1-4 are 21 days)
  For the primary parameters to be assessed on the resected melanoma an objective scoring system will be established by a pathologist, grading each specimen with a score of 0, +, ++, +++. Changes in number of Necrotic Tumor Cells from baseline will be evaluated using a paired McNemar's test for binary outcomes. Quantitative assessment of necrosis of tumor cells will be measured and scored with a value ranging from 0% - 100% of tumor area.
Histological Parameters: Change in Apoptosis from Baseline | Baseline, Cycle 1, Cycle 2, Cycle 4 (cycle length is 21 days)
  For the primary parameters to be assessed on the resected melanoma an objective scoring system will be established by a pathologist, grading each specimen with a score of 0, +, ++, +++.
Histological Parameters: Change in Inflammatory Infiltrate in the tumor from Baseline | Baseline, Cycle 1, Cycle 2, Cycle 4 (cycle length is 21 days)
  For the primary parameters to be assessed on the resected melanoma an objective scoring system will be established by a pathologist, grading each specimen with a score of 0, +, ++, +++.
Histological Parameters: Change in Cellular Phenotype of Infiltrate | Baseline, Cycle 1, Cycle 2, Cycle 4 (cycle length is 21 days)
  Cellular phenotype of infiltrate within the tumor will be summarized by descriptive statistics. Changes from baseline will be evaluated using a paired McNemar's test for binary outcomes.
Histological Parameters: Change in hu14.18-IL2 in the tumor from Baseline | Baseline, Cycle 1, Cycle 2, Cycle 4 (cycle length is 21 days)
  Presence hu14.18-IL2 within the tumor will be summarized by descriptive statistics. Changes from baseline will be evaluated using a paired McNemar's test for binary outcomes.
Pharmacokinetic (PK) Parameters: alpha half-life | At baseline, course 1 day 5, and day 5 of courses 2 & 4 (cycle length is 21 days)
  Pharmacokinetic assessments will be performed on multiple serum specimens for each subject. The analysis of all PK parameters will be performed using the PK analysis population. The distribution half-life called alpha half-life (t1/2 alpha) will be summarized by dose level with simple summary statistics.
Pharmacokinetic (PK) Parameters: beta half-life | At baseline, course 1 day 5, and day 5 of courses 2 & 4 (cycle length is 21 days)
  Pharmacokinetic assessments will be performed on multiple serum specimens for each subject. The analysis of all PK parameters will be performed using the PK analysis population. The elimination half-life called beta half-life (t1/2 beta) will be summarized by dose level with simple summary statistics.
Pharmacokinetic (PK) Parameters: Area Under the Curve (AUC) | At baseline, course 1 day 5, and day 5 of courses 2 & 4 (cycle length is 21 days)
  Pharmacokinetic assessments will be performed on multiple serum specimens for each subject. The analysis of all PK parameters will be performed using the PK analysis population. AUC will be summarized by dose level with simple summary statistics.
Pharmacokinetic Parameters: Clearance (CL) | At baseline, course 1 day 5, and day 5 of courses 2 & 4 (cycle length is 21 days)
  Pharmacokinetic assessments will be performed on multiple serum specimens for each subject. The analysis of all PK parameters will be performed using the PK analysis population. Clearance will be summarized by dose level with simple summary statistics.
Pharmacokinetic (PK) Parameters: Relationship between Dose and AUC | At baseline, course 1 day 5, and day 5 of courses 2 & 4 (cycle length is 21 days)
  Scatterplots will be used to explore possible associations between the dose and area under the curve (AUC). The Jonckheere-Terpstra trend test will be performed to determine the significance of the association between increasing dose level and AUC.
Pharmacokinetic (PK) Parameters: Relationship PK parameters and Toxicity | At baseline, course 1 day 5, and day 5 of courses 2 & 4 (cycle length is 21 days)
  Logistic regression analyses will be performed to correlate PK parameters with toxicity (grade >= 3 vs. grade 0-2) and response.

OTHER OUTCOMES:
Analysis of Antibody Resistance: OR | Up to 5 years
  Clinical outcomes such as OR, duration of response, CB, PFS, and OS will be analyzed separately among subjects who were resistant to prior treatment with anti-CTLA-4 and/or anti-PD1/PD-L1 antibodies and those who lacked resistance in a subgroup analysis. This comparison is by necessity exploratory in nature and hypothesis generating.
Analysis of Antibody Resistance: Duration of Response | Up to 5 years
  Clinical outcomes such as OR, duration of response, CB, PFS, and OS will be analyzed separately among subjects who were resistant to prior treatment with anti-CTLA-4 and/or anti-PD1/PD-L1 antibodies and those who lacked resistance in a subgroup analysis. This comparison is by necessity exploratory in nature and hypothesis generating.
Analysis of Antibody Resistance: CB | Up to 5 years
  Clinical outcomes such as OR, duration of response, CB, PFS, and OS will be analyzed separately among subjects who were resistant to prior treatment with anti-CTLA-4 and/or anti-PD1/PD-L1 antibodies and those who lacked resistance in a subgroup analysis. This comparison is by necessity exploratory in nature and hypothesis generating.
Analysis of Antibody Resistance: PFS | Up to 5 years
  Clinical outcomes such as OR, duration of response, CB, PFS, and OS will be analyzed separately among subjects who were resistant to prior treatment with anti-CTLA-4 and/or anti-PD1/PD-L1 antibodies and those who lacked resistance in a subgroup analysis. This comparison is by necessity exploratory in nature and hypothesis generating.
Analysis of Antibody Resistance: OS | Up to 5 years
  Clinical outcomes such as OR, duration of response, CB, PFS, and OS will be analyzed separately among subjects who were resistant to prior treatment with anti-CTLA-4 and/or anti-PD1/PD-L1 antibodies and those who lacked resistance in a subgroup analysis. This comparison is by necessity exploratory in nature and hypothesis generating.
Analysis of GD2+ vs GD2- Patients: OR | Up to 5 years
  Clinical outcomes such as OR, duration of response, CB, PFS and OS and treatment associated selected biologic effects will be analyzed separately among patients who are GD2+ and those who are GD2- in a subgroup analysis. These outcome measures will be compared using two-sample t-test, log rank test and chi-square/Fisher's exact test between the two groups of patients who are GD2+ and who are GD2-.
Analysis of GD2+ vs GD2- Patients: Duration of Response | Up to 5 years
  Clinical outcomes such as OR, duration of response, CB, PFS and OS and treatment associated selected biologic effects will be analyzed separately among patients who are GD2+ and those who are GD2- in a subgroup analysis. These outcome measures will be compared using two-sample t-test, log rank test and chi-square/Fisher's exact test between the two groups of patients who are GD2+ and who are GD2-.
Analysis of GD2+ vs GD2- Patients: CB | Up to 5 years
  Clinical outcomes such as OR, duration of response, CB, PFS and OS and treatment associated selected biologic effects will be analyzed separately among patients who are GD2+ and those who are GD2- in a subgroup analysis. These outcome measures will be compared using two-sample t-test, log rank test and chi-square/Fisher's exact test between the two groups of patients who are GD2+ and who are GD2-.
Analysis of GD2+ vs GD2- Patients: PFS | Up to 5 years
  Clinical outcomes such as OR, duration of response, CB, PFS and OS and treatment associated selected biologic effects will be analyzed separately among patients who are GD2+ and those who are GD2- in a subgroup analysis. These outcome measures will be compared using two-sample t-test, log rank test and chi-square/Fisher's exact test between the two groups of patients who are GD2+ and who are GD2-.
Analysis of GD2+ vs GD2- Patients: OS | Up to 5 years
  Clinical outcomes such as OR, duration of response, CB, PFS and OS and treatment associated selected biologic effects will be analyzed separately among patients who are GD2+ and those who are GD2- in a subgroup analysis. These outcome measures will be compared using two-sample t-test, log rank test and chi-square/Fisher's exact test between the two groups of patients who are GD2+ and who are GD2-.
PD-L1 expression | up to 5 years
  PD-L1 expression level will be compared between baseline and after initiation of treatment using linear mixed effects model after suitable transformation of PD-L1 expression level. Clinical outcomes such as OR, duration of response, CB, PFS and OS and treatment associated selected biologic effects will be analyzed separately among patients who are PDL1+ and those who are PD-L1- in a subgroup analysis. In addition, these outcome measures will be compared using two-sample t-test, log rank test and chi-square/Fisher's exact test between the two groups of patients who are PD-L1+ and who are PD-L1-.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sondel, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Mark R Albertini, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/